CLINICAL TRIAL: NCT01275859
Title: Neoadjuvant Letrozole and Lapatinib in Postmenopausal Women With ER and Her2 Positive Breast Cancer
Brief Title: Neoadjuvant Combined Endocrine and HER2 Target Therapy in Postmenopausal Women With ER and Her2 Positive Breast Cancer
Acronym: Neo-All-In
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Bae Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0729
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant; Letrozole; Lapatinib; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole, Lapatinib (Experimental): Letrozole 2.5mg po qd + Lapatinib 1500mg po qd for 18-21 wks
  Interventions: Drug: Letrozole, Lapatinib

INTERVENTIONS:
Drug: Letrozole, Lapatinib — Letrozole 2.5mg po qd+ Lapatinib 1500mg po qd for 18-21 wks
  Other Names: Femara; Tykerb

SUMMARY:
Cross-talk between epidermal growth factors and the ER occurs at multiple levels and seems to play a crucial role in breast cancer progression and endocrine resistance.Combined HER1/HER2-targeted therapy with aromatase inhibitors for ER-positive and HER-2 positive postmenopausal breast cancer might enhance response and block emergence of endocrine resistant tumor.

DETAILED DESCRIPTION:
1. To evaluate the efficacy of the neoadjuvant combination therapy with letrozole and lapatinib in postmenopausal patients with ER-positive and HER2-positive breast cancer.
2. To assess markers predictive of treatment response and outcome in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female patients
* Histologically confirmed invasive breast cancer
* Primary tumor greater than 2cm diameter, measured by sonography
* N0-3 (any N if resectable) and no evidence of distant metastasis (M) (isolated supraclavicular node involvement allowed)
* ER positive (intermediate and strong positive)
* HER2 positive (IHC3+ or FISH positive in case of IHC 2+)
* No evidence of metastasis (M0)
* No prior hormonal, chemotherapy or radiotherapy is allowed
* No breast operation other than biopsy to make diagnosis is allowed
* Postmenopausal women with ECOG Performance Status of 0 or 1
* Postmenopausal, as defined by any of the following:
* At least 55 years of age
* Under 55 years of age and amenorrheic for at least 12 months OR follicle-stimulating hormone (FSH) values ≥ 30 IU/L and estradiol levels ≤ 20 IU/L
* Prior bilateral oophorectomy or prior radiation castration with amenorrhea for at least 6 months
* Adequate hematopoietic, renal, hepatic function:

Exclusion Criteria:

* Patients who received hormonal, chemotherapy or radiotherapy for breast cancer
* Patients who underwent surgery for breast cancer
* Patients with bilateral invasive breast cancer
* Patients with inflammatory breast cancer (T4d)
* Patients without primary tumor (T0) Inability to perform [18F]FES PET imaging due to physical inability, claustrophobia, or other mental illness.
* ER poor disease as defined locally (e.g: Allred score 1-3, H-score<100)
* Patients who have history of cancer other than in situ uterine cervix cancer or non-melanotic skin cancer
* Chronic daily treatment with aspirin (>325mg/day) or clopidogrel (>75mg/day)
* Chronic daily treatment with corticosteroids (dose of >10mg /day ethylprednisolone equivalent)
* Clinically significant cardiovascular disease: CVA/stroke (<6month prior to enroll), MI (<6month prior to enroll), unstable angina, NYHA Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication.
* Hormone replacement therapy within 4 weeks of starting treatment
* Known hypersensitivity to any of the study drugs including ditosylate monohydrate salt
* Pregnant or nursing mother (if applicable)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
pCR | 2010 Nov- 2012 May
  To evaluate the pathologic complete response (pCR) rate to lapatinib combined with letrozole in neoadjuvant setting

SECONDARY OUTCOMES:
SUV for [18F]FES PET | 2010 Nov- 2012 May
  * To evaluate clinical overall response (cORR) rate, disease free survival (DFS), overall survival (OS)
  * To assess tolerability and QOL
  * To assess MRI response rate
  * To identify biological predictors of response to lapatinib combined letrozole treatment
  * To determine the correlation of [18F]FES PET with biological and imaging predictors of response to the combined modalities
  * To evaluate the diagnostic value of SUV for [18F]FES PET in the prediction of pathologic, clinical response to neoadjuvant HER2 target- and endocrine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Nedical Center, Seoul, South Korea